CLINICAL TRIAL: NCT06468241
Title: The Effect of Listening to Music and Progressive Relaxation Exercise on Fatigue and Sleep in Multiple Sclerosis: A Randomized Controlled Study
Brief Title: The Effect of Music and Progressive Relaxation Exercise on Fatigue and Sleep in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ahsen Taştan Gürkan, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU-AHSENTASTANGURKAN-001
Record Dates: First submitted 2023-08-01; First posted 2024-06-21 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Fatigue; Sleep
Keywords: Multiple Sclerosis; Progressive relaxation exercise; listening to music; sleep; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive relaxation exercise group (Experimental): progressive relaxation exercise intervention and measurement with scales and wearable technology
  Interventions: Other: Progressive relaxation exercise
- Music group (Experimental): music listening intervention and measurement with scales and wearable technology
  Interventions: Other: Listening to music
- Control group (No Intervention): No intervention and measurement with scales and wearable technology

INTERVENTIONS:
Other: Progressive relaxation exercise — For the progressive relaxation exercise group, a progressive relaxation exercise session will be applied to the participants 3 times a week for four weeks.
  Arms: Progressive relaxation exercise group
Other: Listening to music — For the music listening group, the participants will listen to the Turkish music makams ("uşşak" and "rast") three times a week for four weeks.
  Arms: Music group

SUMMARY:
Multiple Sclerosis (MS) is a chronic complex neurodegenerative disease that targets the central nervous system and is autoimmune. The prevalence of fatigue in individuals diagnosed with MS varies between 50% and 81%. It is one of the most common, disabling and complex symptoms of MS. Another common symptom in MS patients is sleep problems. Sleep problems are seen in approximately 70% of MS patients. Non-pharmacological interventions have been used in recent years for the management of fatigue and sleep problems in MS. The effects of Progressive relaxation exercises (PGE), one of the non-pharmacological methods, on sleep and fatigue symptoms in MS patients have been reported. It has been reported that the implementation of progressive relaxation exercises in MS is a supportive intervention for sleep quality and fatigue and is recommended for future research.

Another initiative that is planned to be used within the scope of this research proposal is listening to music. Although rhythm and music have recently become a topic of interest in the field of neurological rehabilitation, their value in practice has not yet been fully discovered. Suggestions are given to objectively define sleep disorders in MS and to focus on this symptom of MS. It has been determined that music shows promise in improving sleep, but more research is needed on improved techniques for sleep measurement.

The main purpose of this research is to reveal the effects of listening to music and progressive relaxation exercise on fatigue and sleep in Multiple Sclerosis. The research was planned as a randomized controlled experimental study in a three-measure design with three groups (music listening, progressive relaxation exercise, and control group). The sample of the project consists of 30 individuals with MS diagnosis and meeting the inclusion criteria. In data collection, it is planned to use of the Introductory Information Form, which includes the sociodemographic characteristics of the patients, the characteristics of the disease and sleep habits, the Fatigue Severity Scale, the Fatigue Impact Scale and the Pittsburgh Sleep Quality Index and wearable technology. Data were analysed with Statistical Package for the Social Sciences (SPSS) V23 and R software. In addition to descriptive analyses, In addition to descriptive analyses, multiple comparisons by group and time were performed using generalised linear model analyses.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic complex neurodegenerative disease that targets the central nervous system and is autoimmune. The prevalence of fatigue in individuals diagnosed with MS varies between 50% and 81%. It is one of the most common, disabling and complex symptoms of MS. Another common symptom in MS patients is sleep problems. Sleep problems are seen in approximately 70% of MS patients. It has been reported that sleep disorders affect the course of MS negatively. Non-pharmacological interventions have been used in recent years for the management of fatigue and sleep problems in MS. The effects of Progressive relaxation exercises (PGE), one of the non-pharmacological methods, on sleep and fatigue symptoms in MS patients have been reported. It has been reported that the implementation of progressive relaxation exercises in MS is a supportive intervention for sleep quality and fatigue and is recommended for future research.

Another initiative that is planned to be used within the scope of this research proposal is listening to music. Although rhythm and music have recently become a topic of interest in the field of neurological rehabilitation, their value in practice has not yet been fully discovered. Suggestions are given to objectively define sleep disorders in MS and to focus on this symptom of MS. It has been determined that music shows promise in improving sleep, but more research is needed on improved techniques for sleep measurement.

Polysomnography (PSG) is used for the objective measurement of sleep. However, it may cause poorer quality sleep as it requires participants to sleep in a laboratory environment. For this reason, it is important to use objective measurement tools that patients can do in their own environment.

The main purpose of this research is to reveal the effects of listening to music and progressive relaxation exercise on fatigue and sleep in Multiple Sclerosis. The research was planned as a randomized controlled experimental study in a three-measure design with three groups (music listening, progressive relaxation exercise, and control group). The sample of the project consists of 30 individuals with MS diagnosis and meeting the inclusion criteria. In data collection, it is planned to use of the Introductory Information Form, which includes the sociodemographic characteristics of the patients, the characteristics of the disease and sleep habits, the Fatigue Severity Scale, the Fatigue Impact Scale and the Pittsburgh Sleep Quality Index and wearable technology. Data were analysed with Statistical Package for the Social Sciences (SPSS) V23 and R software. In addition to descriptive analyses, In addition to descriptive analyses, multiple comparisons by group and time were performed using generalised linear model analyses.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having a diagnosis of MS for at least six months and being in remission
* To be between 0-3.5 points on the Expanded Disability Status Scale (EDSS),
* Having the disease type Relapsing Remitting (RRMS),
* Having a score of 4 or more on the Fatigue Severity Scale, (In the Fatigue Severity Scale, 4 points is the cut-off value and scores of 4 and above indicate pathological fatigue.)
* Having a score above 5 on the Pittsburgh Sleep Quality Index, (A total score of >5 indicates that the sleep quality of the individual is inadequate.)
* To be residing in "Samsun,Turkey",
* Having the ability to use technology with computer/phone and internet facilities,
* To voluntarily accept participation in research.

Exclusion Criteria:

* Having a chronic disease other than MS,
* Having a sleep disorder diagnosed for different reasons,
* To be diagnosed with a psychiatric disorder that may prevent obtaining a healthy result from the study and affect sleep (Major depressive disorder, serious anxiety disorders, severe psychiatric conditions, etc.),
* Using a regular non-pharmacological method (Yoga, psychotherapy, etc.) for sleep and fatigue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The effect of progressive relaxation exercise and listening to music on sleep quality | two and four weeks after starting the intervention
  It will be measured with the Pittsburgh Sleep Quality Index
The effect of progressive relaxation exercise and listening to music on fatigue | two and four weeks after starting the intervention
  It will be measured with the Fatigue Severity Scale
The effect of progressive relaxation exercise and listening to music on fatigue effect | two and four weeks after starting the intervention
  It will be measured with the Fatigue Impact Scale
The effect of progressive relaxation exercise and listening to music on sleep | two and four weeks after starting the intervention
  It will be measured with the Wearable Tecnology

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)